CLINICAL TRIAL: NCT02900521
Title: The Brest Registry of Stroke
Brief Title: Population-based Brest Stroke Registry
Acronym: BREST
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Collaborators: Santé publique France-InVS (Institut National de Veille sanitaire) (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: REGISTRE AVC
Record Dates: First submitted 2016-08-22; First posted 2016-09-14 (Estimated); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Cerebral (CVAs); Ischemic Cerebrovascular Accident; Stroke; Brain Ischemia; Brain Hemorrhage; Ischemic Stroke; Hemorrhagic Stroke; Cerebrovascular Disorders; Transient Ischemic Attack (TIA)
MeSH Terms: conditions — Ischemic Stroke; Stroke; Brain Ischemia; Intracranial Hemorrhages; Hemorrhagic Stroke; Cerebrovascular Disorders; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The registry is the main objective exhaustive list of cases validated stroke brain on a geographical area defined to calculate an incidence.

DETAILED DESCRIPTION:
The main objective of Brest Stroke Registry is to regroup all confirmed cases of stroke over a defined geographical zone in order to calculate an incidence.

There are three prospective medium-term goals:

- In respect with public health epidemiology:

1. To obtain incidence data and evaluate the regional and international divergences
2. To obtain the mortality data in short and long term. Since the onset of the registry, it has been implemented a study on the mortality of stroke patients of Brest Registry. This study has been realized independently for both types of stroke, i.e. ischemic and hemorrhagic, with different caused mortality. This mortality was studied at medium-term (≤ 28 days) as well as at long-term (> 28 days). There will be a collaboration project between Public Health Surveillance (InVS), Brest University Hospital and Rennes network on all causes of death.
3. Pharmaco-epidemiology

In clinical terms, the registry offers an opportunity to do an inventory of all current practices (diagnosis, therapies and the subsidiaries) and propose in this manner the best management of stroke. This strategy is in line with the pilot programs deployed by the French High Health Authority (HAS) for improvement of quality and safety of the health care. The bleeding risk associated with anticoagulants and anti-platelet agents in people of Brest as well as that of Dijon and Lille (in collaboration with their respective registry) will be analyzed.

This study has gained a particular characteristic since 2012 with emerging new oral anticoagulants (OAC) which have shown less associated bleeding risks compared with vitamin K antagonists (randomized controlled trials).

•In terms of clinical research :

1. Study the impacted consequences of stroke by socio-economic characteristics of the territories in the Pays de Brest
2. Identify short and long term clinical predictors of mortality in patients who have had a hemorrhagic stroke.
3. To identify clinical predictors of mortality in the short and long-term patients with ischemic stroke.
4. To identify genetic predictors of mortality and long-term recurrence of patients with ischemic stroke
5. Identify stroke identification algorithm from existing databases

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic validated for one of the following pathologies:
* Ischemic stroke,
* Non-traumatic intracranial hematoma
* Cerebral venous thrombosis Diagnostic after December 31, 2007 Age > 15 years on the date of the diagnostic Patient domiciled at the time of the diagnostic in one of the 79 communes defined beforehand

Exclusion Criteria:

* Age ≤ 15 years
* Validated diagnosis (see below, § 4.2.2) of aneurysmal subarachnoid hemorrhage cerebrovascular
* Diagnosis made before 1 January 2008
* Unconfirmed diagnosis
* Patient domiciled outside the previously defined area of residence

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnostic validated for one of the following pathologies:
  * Ischemic stroke,
  * Non-traumatic intracranial hematoma
  * Cerebral venous thrombosis Diagnostic after December 31, 2007 Age > 15 years on the date of the diagnostic Patient domiciled at the time of the diagnostic in one of the 79 communes defined beforehand
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2008-01 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Type of stroke (ischemic or haemorrhagic) | Inclusion
  The type of stroke ischemic or haemorrhagic will be collected from physician diagnostic

SECONDARY OUTCOMES:
Patient outcome | Every year after the inclusion during 10 years
  Patient outcome (mortality) wanted by mail from towns of birth

CONTACTS AND LOCATIONS:
Overall Officials: Serge TIMSIT, Principal Investigator — CHRU La Cavale Blanche - BREST - FRANCE
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes